CLINICAL TRIAL: NCT01777906
Title: Comparison of Topical Nasal Steroids in Postoperative Sinus Patients With Nasal Polyps
Brief Title: Study of the Efficacy of Topical Nasal Steroids Patients With Nasal Polyps
Acronym: dexamethasone
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Kristin Seiberling, MD, Principil investigator, Loma Linda University
Other Study IDs: 5130043
Record Dates: First submitted 2013-01-24; First posted 2013-01-29 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Size of Nasal Polyps; Control of Symptoms
Keywords: nasal polyps; nasal steriod sprays
MeSH Terms: conditions — Nasal Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Fluticasone: Fluticasone nasal spray will be given 2 sprays twice a day for 6 weeks.
- Dexamethasone sodium phosphate 0.032%: Dexamethasone 0.032% nasal spray will be given at a dose of 2 sprays twice a day for 6 weeks.

SUMMARY:
Topical nasal steroid sprays are the mainstream treatment for patients with nasal polyps. Polyps tend to recur after surgery and topical nasal steroid sprays are used as the primary medical management to prevent continued growth. More recently high dose topical nasal steroid sprays are used. It is thought that the higher dose will penetrate the sinus cavities at an increased dose and will allow for greater control of polyp growth. Safety studies have been performed which have shown no suppression of the pituitary axis with long term high dose topical steroid or changes in intraocular pressure. However, studies in efficacy are limited despite their widespread use. The objective of this study will be to compare the effectiveness of two topical nasal steroid sprays in patients with recurrent nasal polyps.

DETAILED DESCRIPTION:
Recruitment plan- Patients with nasal polyps who have had sinus surgery at least 3 months prior and documented nasal polyps by endoscopy will be prospectively recruited. This will be a randomized blinded study. Patients will be randomized into two groups- group 1 will received topical fluticasone and group 2 will receive topical dexamethasone spray to the nasal cavity. The investigator will be blinded as to which group the subjects are placed in. The medications will be given out from the inland compounding pharmacy located at 24747 Redlands Blvd, in Loma Linda.

Procedures

1. At the time of enrollment nasal endoscopy will be performed to confirm the diagnosis of nasal polyps and to grade the size of the polyps. Polyp size will be graded by the following scale: 0- no polyps, 1- polypoid mucosa, 2- polyps within sinus not occluding ostium, 3- polyps occluding ostium filling nasal cavity
2. Subjects will be asked to fill out a SNOT 20 survey before the start of therapy.
3. Subjects will be randomized into 2 groups by the flip of a coin. The investigator will be blinded to which group the subject is placed in. The pharmacist (Raylene Mote, Inland compounding pharmacy) who compounds the medications will be the only one aware of which medication was given.
4. Subjects will pick up their medication at the inland compounding pharmacy and will be instructed to use the nasal spray- 2 sprays twice a day for 6 weeks.
5. After 6 weeks the subjects will return to the office for repeat nasal endoscopy and will be asked to fill out a SNOT 20 survey.
6. Continued therapy of the nasal steroid spray will be at the discretion of the physician. If subjects do not appear to be responding the nasal steroid spray the medication will be altered as deemed medically necessary.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with nasal polyps who have had sinus surgery at least 3 months prior to enrollment.

Exclusion Criteria:

* Allergy to steroids
* Glaucoma
* Cataracts

Ages: 17 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Group 1 - will be given fluticasone nasal spray Group 2- will be given dexamethasone nasal spray The 2 groups will be compared in terms of symptom control and polyp size
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Comparison of topical nasal steroids in postoperative sinus patients | 1 year
  Primary outcome will be symptomatic improvement measured by the SNOT 20 survey and physical size of polyps as measured by nasal endoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Seiberling, MD, Principal Investigator — Loma Linda University
Locations (1):
- Sinus and Allergy Center, Loma Linda, California, United States